CLINICAL TRIAL: NCT01777204
Title: Non-invasive Assessment of Gastrointestinal Transit and Motility in Renal Transplant Recipients Employing a Biomagnetic Technique
Brief Title: Gastrointestinal Transit and Motility in Renal Transplant Recipients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade Estadual de Ciências da Saúde de Alagoas (Other)
Collaborators: UPECLIN HC FM Botucatu Unesp (Other); University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Maria do Carmo Borges, Doctor, Universidade Estadual de Ciências da Saúde de Alagoas
Other Study IDs: FAPEAL-20110714-TX
Record Dates: First submitted 2013-01-23; First posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Change of Transit or Circulation; Effects of Immunosuppressant Therapy
Keywords: Renal transplant, Gastrointestinal motility, Biomagnetism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (7):
- Tacrolimus: Influence of tacrolimus on gastrointestinal transit and motility in renal transplant recipients.
- Cyclosporine: Influence of cyclosporine on gastrointestinal transit and motility in renal transplant recipients.
- Mycophenolate mofetil: Influence of mycophenolate mofetil on gastrointestinal transit and motility in renal transplant recipients.
- Mycophenolate sodium: Influence of mycophenolate sodium on gastrointestinal transit and motility in renal transplant recipients.
- Everolimus: Influence of everolimus on gastrointestinal transit and motility in renal transplant recipients.
- Sirolimus: influence of sirolimus on gastrointestinal transit and motility in renal transplant recipients.
- Without immunosuppression: Gastrointestinal transit and motility in healthy volunteers.

SUMMARY:
Gastrointestinal (GI) complications after renal transplantation are commonly reported as side effects of immunosuppressive agents. Despite this, motility disorders have been scantily studied. Alternating Current Biosusceptometry (ACB) are biomagnetic sensors designed for a wide range of applications. In clinical practice, their non-invasive and radiation free features provide an excellent approach for monitoring of GI transit as alternative to scintigraphy and breath tests. The aim of this study is to examine GI transit and motility of solids in stable renal transplant recipients to determine the potential influence of immunosuppressive therapy on gastrointestinal parameters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteer or Renal Transplant Patients
* Signed informed consent obtained
* Fasted since midnight

Exclusion Criteria:

* Subject has known GI related symptoms complaints or GI diseases
* Subject has cancer or other life threatening diseases or conditions
* Subject is pregnant
* Subject has undergone abdominal surgery
* Drug abuse or alcoholism
* Subject has cardiac pacemaker
* Subject takes any medication affecting GI motility

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Renal transplant recipients from Alagoas, Brazil
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Influence of tacrolimus and cyclosporine on gastrointestinal transit | one year

CONTACTS AND LOCATIONS:
Overall Officials: Maria do Carmo B Teixeira, Dr, Principal Investigator — Universidade Estadual de Ciências da Saúde de Alagoas
Locations (1):
- Universidade Estadual de Ciências da Saúde de Alagoas, Maceió, Alagoas, Brazil